CLINICAL TRIAL: NCT04730635
Title: A Clinical Study to Evaluate a Cognitive Platform to Support Development of Symptomatic Therapies in Participants at Risk for Alzheimer's Disease
Brief Title: Cognition Platform Study in Participants at Risk for Alzheimer's Disease (AD) (MK-0000-413)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0000-413; MK-0000-413 (Other: Merck)
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Single-blind (placebo run-in) followed by double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donepezil (Experimental): Participants receive donepezil in doses up to 10 mg once daily (QD), orally in a scheduled titration for Days 1-56. The total treatment duration is 56 days.
  Interventions: Drug: Donepezil
- Placebo (Placebo Comparator): Participants receive placebo QD, orally for Days 1-56. The total treatment duration is 56 Days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donepezil — Donepezil 5 mg capsules for a total daily dose of up to 10 mg QD, orally, for Days 1-56.
  Other Names: MK-0000; Donepezil hydrochloride; Aricept
  Arms: Donepezil
Drug: Placebo — Dose matched placebo capsule QD, orally for Days 1-56.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the ability of a repeated high-frequency site-based computerized cognitive assessment to evaluate the potential treatment effects of donepezil (MK-0000) compared with placebo among participants with mild cognitive impairment (MCI) or mild Alzheimer's Disease (AD). The primary study hypothesis is that the average percentage of correct responses on one card learning (OCL) task will be ≥2 percentage points in participants receiving donepezil compared with participants receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Has an Mini Mental State Examination (MMSE) score between 18 and 28 (inclusive) at Screening (Visit 1) and Baseline (Visit 2)
* Has a diagnosis of mild cognitive impairment (MCI) or mild Alzheimer's Disease (AD)
* Has an Modified Hachinski Ischemia Scale (MHIS) score of ≤4
* Must have a reliable and competent study partner/informant who accompanies participant to study visits and participates in assessments
* Be willing to provide a blood sample for Apolipoprotein E (APOE) genotyping
* Does not have intellectual disability
* Be able to speak, read, hear, and understand the language of the study staff and the Informed Consent Form (ICF)
* Be able and willing to adhere to the study visit schedule
* Have visual acuity, visual function, hearing, and gross and fine motor skills adequate to support study participation
* Be capable of performing the Cogstate battery assessments, as demonstrated at the Baseline/Familiarization Visit (Visit 2)
* A female participant is eligible to participate if she is a woman of nonchildbearing potential (WONCBP)

Exclusion Criteria:

* Is at imminent risk of self-harm
* Has evidence of a clinically relevant neurological disorder other than AD at screening, including but not limited to: Parkinson's disease, frontotemporal dementia, Huntington's disease, amyotrophic lateral sclerosis, multiple sclerosis, progressive supranuclear palsy, dementia with Lewy bodies, other types of dementia, neurosyphilis or that led to persistent cognitive deficits, or has a history of seizures or epilepsy within the last 5 years before screening
* Has a known history of stroke or has a diagnosis of vascular dementia
* Has history of multiple episodes of head trauma, or head trauma resulting in protracted loss of consciousness, or serious infectious disease affecting the brain, within the prior 3-5 years
* Has evidence of a clinically relevant or unstable psychiatric disorder, based on Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5), including schizophrenia or other psychotic disorder, bipolar disorder, major depression, or delirium
* Has a recent or ongoing, uncontrolled, clinically significant medical condition within 2 months of the Screening visit
* Has a history of cancer
* Has a relative contraindication to donepezil including sick sinus syndrome, first, second, or third-degree heart block, bradycardia, active gastrointestinal (GI) bleeding, Zollinger-Ellison syndrome, uncontrolled peptic ulcer disease, or uncontrolled asthma
* Has a history of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food. Exception: Participants with selected allergies may be enrolled with Sponsor's approval
* Is positive for Hepatitis B surface antigen (HBsAg), hepatitis C antibodies or human immunodeficiency virus (HIV) [participants with a history of chronic hepatitis C virus with a documented cure and/or a positive serologic test for HCV with a negative HCV viral load may be included]
* Has clinically significant vitamin B12 or folate deficiency in the 6 months immediately before screening, or vitamin B12 or folate deficiency in addition to increased serum homocysteine and methylmalonic acid levels at screening
* Has prior AD treatment
* Has participated in another investigational study within 4 weeks
* Has a known history of structural changes on screening magnetic resonance imaging (MRI) scan that are clinically important, including signs indicative of vascular dementia, large infarct, lacunes in critical areas, space-occupying lesions, or extensive white matter disease
* Is unwilling to or not eligible to undergo a MRI scan (if a prior MRI scan is not available)
* Is pregnant, is attempting to become pregnant, or is nursing children
* Has a history of alcoholism or drug dependency/abuse within the last 5 years prior to the Screening visit
* Consumes greater than 3 glasses of alcoholic beverages per day
* Consumes excessive amounts, defined as greater than 6 servings of coffee, tea, cola, energy drinks, or other caffeinated beverages per day
* Is a regular user of cannabis, any illicit drugs or has a history of drug abuse within approximately 5 years. A participant who is a recreational user of cannabis or other drugs within the past 2 years can be enrolled as long as recreational use does not meet the definition of drug abuse and participant agrees to refrain from substance use for duration of study participation
* Participants must have a negative urine drug screen (UDS) prior to randomization
* Had major surgery within 3 months prior to the Screening visit that would interfere in the participant's ability to fully participate in the study
* Has undergone neuropsychological testing (including the MMSE) or cognitive remediation in the past 4 weeks
* Is or has an immediate family member who is investigational site or Sponsor staff directly involved with this study

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (10):
- United States (8):
  - Collaborative Neuroscience Network ( Site 0010), Long Beach, California
  - Velocity Clinical Research, Hallandale Beach ( Site 0013), Hallandale, Florida
  - Charter Research - Lady Lake ( Site 0025), Lady Lake, Florida
  - iResearch Atlanta ( Site 0005), Decatur, Georgia
  - iResearch Savannah ( Site 0023), Savannah, Georgia
  - Pennington Biomedical Research Center ( Site 0006), Baton Rouge, Louisiana
  - Insight Clinical Trials ( Site 0020), Beachwood, Ohio
  - North Texas Clinical Trials - Fort Worth - West Rosedale ( Site 0022), Fort Worth, Texas
- Australia (2):
  - Royal Adelaide Hospital-CALHN Memory Trials ( Site 0031), Adelaide, South Australia
  - Austin Health ( Site 0030), Heidelberg, Victoria

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment-naïve male and female participants with mild cognitive impairment (MCI) or mild Alzheimer's Disease (AD) between the ages of 55 and 85 years (inclusive) will be enrolled in this trial.
Period: Overall Study
Arm/Group | Donepezil | Placebo
Started | 29 | 15
Completed | 28 | 14
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil | Placebo | Total
Number analyzed (Participants) | 29 | 15 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.3 (7.6) | 68.4 (7.7) | 68.4 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 12 | 3 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 19
  Not Hispanic or Latino | 17 | 8 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 19 | 9 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Averaged Correct Response Rate on the One Card Learning Task to Week 8
Description: One Card Learning (OCL) uses a pattern separation paradigm to assess visual memory. The change from baseline of correct responses on the OCL task up to Week 8 is compared in participants receiving donepezil with participants receiving placebo. Change from baseline was the averaged correct response rate at Week 8 minus the correct response rate at baseline.
Time Frame: Baseline, Up to Week 8
Population: All participants who received at least one dose of study medication and yielded at least one measurement for that outcome measure.
Measure: Mean (Standard Deviation); unit: Proportion of correct response
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 23 | 13
Proportion of correct response | 0.055 (0.078) | 0.034 (0.091)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; There was a threshold of ≥2 percentage points. A posterior probability value >55% was required to satisfy the primary hypothesis; Test type: Other; Posterior Probability = 46.30

2. Secondary Outcome: Change From Baseline in Standard Deviation for Averaged Correct Response Rate on the OCL Task (Arcsine Square Root Transformed) to Week 8
Description: OCL uses a pattern separation paradigm to assess visual memory. Change in standard deviation from baseline for correct response rate on the OCL task up to Week 8 is compared in participants with mild cognitive impairment (MCI) or mild Alzheimer's Disease (AD) receiving donepezil with participants receiving placebo. Change from baseline was the standard deviation for correct response rate at Week 8 minus the standard deviation for correct response rate at baseline. Standard deviations are reported in arcsine square root (sqrt) transformed correct response (CR) rate.
Time Frame: Baseline, Up to Week 8
Population: as for outcome 1
Measure: Number; unit: Arcsine sqrt transformed proportion CR
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 23 | 13
Arcsine sqrt transformed proportion CR
  MCI: number analyzed (Participants) | 16 | 9
  MCI | 0.078 | 0.074
  Mild AD: number analyzed (Participants) | 7 | 4
  Mild AD | 0.080 | 0.097
Statistical Analysis 1: Comparison: Donepezil; There was a threshold of ≤ 0.1 for this standard deviation change. A posterior probability value >70% was required to satisfy this secondary hypothesis; Test type: Other; Posterior Probability = 80.67

3. Secondary Outcome: Change From Baseline in Averaged Correct Response Rate on the OCL Task to Week 8 in Participants Receiving Donepezil
Description: OCL uses a pattern separation paradigm to assess visual memory. The change from baseline of correct responses on the OCL task up to Week 8 in participants receiving donepezil is presented. Change from baseline was the averaged correct response rate at Week 8 minus the correct response rate at baseline. Per protocol, the placebo group was not included in this analysis.
Time Frame: Baseline, Up to Week 8
Population: All participants who received at least one dose of donepezil and yielded at least one measurement for that outcome measure. Per protocol, the placebo group was not included in this analysis.
Measure: Mean (Standard Deviation); unit: Proportion of correct response
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 23 | 0
Proportion of correct response | 0.055 (0.078) |
Statistical Analysis 1: Comparison: Donepezil; Test type: Other; Posterior Probability = 98.8

ADVERSE EVENTS:
Time Frame: Up to Week 10 (up to 70 days)
Description: All-Cause Mortality (ACM) was reported for all randomized participants.
  Serious AEs and Other AEs were reported for the Safety Population: all randomized participants who received at least 1 dose of study medication.
Arm/Group | Donepezil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/15
Other Adverse Events (participants affected / at risk) | 16/29 | 4/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=29) | Placebo (N=15)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=29) | Placebo (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 3 (3) | 0 (0)
Emotional distress (Psychiatric disorders) | 1 (1) | 0 (0)
Hypnagogic hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT04730635/Prot_SAP_000.pdf